CLINICAL TRIAL: NCT04035070
Title: Effect of Irrigation With Antibiotic-containing Solutions Versus Sodium Hypochlorite on Postoperative Pain and Intra-canal Bacteria in Teeth With Necrotic Pulps (a Randomized Double-blind Clinical Trial)
Brief Title: Effect of Irrigation With Antibiotic-containing Solutions on Postoperative Pain and Intra-canal Bacteria
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Michel Karam Eissa Elias, Assistant lecturer at endodontic department - School of dentistry - New Giza University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBC-CU-2019-10-145
Record Dates: First submitted 2019-07-21; First posted 2019-07-29 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Necrotic Pulp
Keywords: antibiotic-containg solution; co-amoxiclav-clindamycin solution; MTAD; sodium hypochlorite; postoperative pain; antimicrobial efficacy; root canal irrigation
MeSH Terms: conditions — Dental Pulp Necrosis; Pain, Postoperative | interventions — MTAD (intracanal irrigant); Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Root canal irrigation with co-amoxiclav-clindamycin solution (Experimental): Alternate irrigation with 1 mL antibiotic-containing solution followed by 4 mL 2.5% sodium hypochlorite solution between each size instrument and the consequent one. The antibiotic-containing solution will be prepared by mixing equal quantities of 1.2 gm Co-amoxiclav solution and 600 mg Clindamycin solution at a ratio of 1:1 by volume.
  Interventions: Combination Product: co-amoxiclav-clindamycin solution
- Root canal irrigation with MTAD (Experimental): Irrigation with 5 mL MTAD irrigating solution for 5 minutes between each size instrument and the consequent one.
  Interventions: Combination Product: MTAD
- Root canal irrigation with 2.5% sodium hypochlorite (Active Comparator): Irrigation with 5 mL 2.5% sodium hypochlorite irrigating solution between each size instrument and the consequent one.
  Interventions: Combination Product: 2.5% sodium hypochlorite

INTERVENTIONS:
Combination Product: co-amoxiclav-clindamycin solution — antibiotic-containing solution will be prepared by mixing equal quantities of 1.2gm Co-amoxiclav solution and 600mg Clindamycin solution at a ratio of 1:1 by volume to be used as a root canal irrigating solution
  Arms: Root canal irrigation with co-amoxiclav-clindamycin solution
Combination Product: MTAD — mixture of 3% doxycycline hyclate, 4.25% citric acid and detergent (Tween 80) to be used as a root canal irrigating solution
  Other Names: BioPure MTAD
  Arms: Root canal irrigation with MTAD
Combination Product: 2.5% sodium hypochlorite — It will be prepared by adding 10mL of sterile distilled water to 10mL of 5.25% sodium hypochlorite solution to be used as a root canal irrigating solution
  Arms: Root canal irrigation with 2.5% sodium hypochlorite

SUMMARY:
• The aim of this study is to compare the degree of postoperative pain and the antimicrobial effect in terms of bacterial count reduction after using co-amoxiclav-clindamycin solution versus MTAD and sodium hypochlorite irrigating solutions in patients with necrotic pulp.

DETAILED DESCRIPTION:
* After confirming the diagnosis and making sure that the patient conforms to all eligibility criteria, the principal investigator will enroll the patient in the study.
* The operator will complete treatment of all cases in two visits as follows:

  1. Anesthesia will be achieved using inferior alveolar nerve block for mandibular premolar teeth and infiltration technique for maxillary anterior teeth with local anesthesic solution of 1.8 mL of 2% Mepivacaine HCl with 1:100,000 epinephrine.
  2. Caries and/or coronal restorations will be completely removed with sterile bur and rubber dam will then be applied.
  3. The operative field, including the tooth, the clamp and rubber dam sheet will be cleaned with 30% hydrogen peroxide for 30 seconds, followed by a sterile cotton swab with 5.25% NaOCl for the same period of time and then inactivated with 5% sodium thiosulphate.
  4. Access cavity will be prepared using a sterile round carbide bur size 3 and a sterile Endo-Z bur.
  5. The operative field and the pulp chamber will be cleaned and disinfected once again in the same way mentioned above.
  6. Patency of the root canals will be achieved using #10 or #15 size stainless steel hand K-files. Working length (WL) will be determined using an electronic apex locator then confirmed radiographically to be 1 mm shorter than radiographic apex.
  7. Debridement and mechanical preparation will be performed with the initial file along with 2 mL of 0.9% sterile saline solution and then a pre-instrumentation sample will be collected from the root canal.
  8. The pre-instrumentation sample (S1) will be collected as follows: a sterile paper point will be placed inside the root canal to soak up the fluid in the canal to a level approximately 1 mm short of the tooth apex. The paper point will be left in the canal for 60 seconds. This will be repeated using three sterile paper points. Paper points will then be transferred aseptically to tubes containing 20 mL of sterile thioglycolate broth.

     Microbiological analysis To test for the presence of cultivable bacteria, cultures will be inoculated in thioglycolate broth. For the identification of main anaerobic taxa, the root canal samples will be plated on 5% sheep blood agar, neomycin blood agar and phenyl ethyl alcohol agar with metronidazole (5μg, Oxoid, Basingstoke, UK) disc. Cultures will be incubated at 37°C for 72 hours in an anaerobic chamber . In addition, specimens will also be cultured aerobically on 5% sheep blood agar and MacConkey's agar.
  9. Mechanical preparation will be completed in a crown down technique with Protaper Next rotary files set on an endodontic motor adjusted at a speed of 300 rpm and torque of 2 Ncm. In-and-out motions will be applied with stroke lengths not exceeding 3 mm in the cervical, middle, and apical thirds until attaining the established WL. All root canals will be enlarged to size X4 (40.06). The canal will be irrigated and recapitulated after the use of each instrument according to the allocated group as follows:

     Group 1: Alternate irrigation with 1 mL antibiotic-containing solution followed by 4 mL 2.5% sodium hypochlorite solution between each size instrument and the consequent one. The antibiotic-containing solution will be prepared by mixing equal quantities of 1.2 gm Co-amoxiclav solution and 600 mg Clindamycin solution at a ratio of 1:1 by volume.

     Group 2: Irrigation with 5 mL MTAD irrigating solution for 5 minutes between each size instrument and the consequent one.

     Group 3 (control): Irrigation with 5 mL 2.5% sodium hypochlorite irrigating solution between each size instrument and the consequent one.
  10. The root canal will be thoroughly irrigated with the allocated irrigant using a plastic disposable syringe with a gauge 30 side-vented needle reaching 1 mm short of the WL. The canal will then be dried using sterile paper points.
  11. Canals irrigated with NaOCl (groups 1 and 3) will be flushed with 5 mL of 5% sodium thiosulfate to inactivate the NaOCl followed by 5 mL 0.9% sterile saline solution. Canals irrigated with MTAD (group 2) will be flushed with 5 mL 0.9% sterile saline solution.
  12. A post-instrumentation sample (S2) will be taken as previously described and then the cavity will be sealed with a sterile cotton pellet and a temporary filling material .
  13. The patient will be instructed to record their pain level on NRS at 24 and 48 hours postoperatively and will be recalled after 72 hours. The patient will be prescribed Ibuprofen (400 mg) to be taken in case of intolerable pain.
  14. In the recall appointment, the root canal will be accessed under sterile conditions and will be flushed with 1mL sterile saline solution before a third sample (S3) is taken as previously described.
  15. Master cone fit radiograph will be taken and then the root canal will be dried using sterile paper points and filled with gutta percha points and resin-based sealer using cold lateral condensation technique.
  16. Access cavity will be sealed with a temporary filling material and the final restoration will be placed within one week.
  17. The patient will be asked to report any swelling, in such case, he/she will be appointed for clinical examination to assess the severity by a blinded assessor and to determine if systemic antibiotics/drainage will be needed.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary/mandibular single-rooted permanent teeth:

  * Diagnosed clinically with pulp necrosis.
  * Absence of spontaneous pain.
  * Normal/slight widening in the periodontal membrane space (PMS).
* Patients' acceptance to participate in the trial.
* Patients who can understand numerical rating scale (NRS) and can sign the informed consent.

Exclusion Criteria:

* Medically compromised patients: Pain levels and healing following treatment would be compromised as these patients show higher incidence of pain and lower healing rate.
* Patients with known allergy to penicillin or penicillin derivatives.
* Pregnant females: Avoid radiation exposure, anesthesia, and medication.
* If analgesics or antibiotics have been administrated by the patient during the past 24 hours preoperatively: Might alter their pain perception.
* Patients reporting bruxism or clenching: Avoid further pressure on an already inflamed tooth inducing subsequent irritation and inflammation.
* Teeth that show association with acute periapical abscess and swelling: Need special treatment steps which could involve additional visits with incision and drainage. Also, it could influence initiation and progression of postoperative pain.
* Greater than grade I mobility or pocket depth greater than 5mm. Need special surgical and/or periodontal therapy.
* Non-restorable teeth.
* Immature teeth.
* Radiographic evidence of periapical radiolucency, external or internal root resorption, vertical root fracture, perforation or calcification.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
postoperative pain: numerical rating scale | up to 48 hours after the first visit
  intensity of pain by numerical rating scale from 0 to 10

SECONDARY OUTCOMES:
intra-canal bacterial count | 72 hours after root canal preparation
  pre and post-instrumentation samples to count intra-canal bacteria (CFU/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Michel K Elias, M.Sc., Principal Investigator — Cairo University; Maged M Negm, Ph.D., Study Director — Cairo University; Heba El-Asfouri, Ph.D., Study Chair — Cairo University
Locations (1):
- Endodontic Department - Faculty of Dentistry - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pak JG, White SN. Pain prevalence and severity before, during, and after root canal treatment: a systematic review. J Endod. 2011 Apr;37(4):429-38. doi: 10.1016/j.joen.2010.12.016. PMID 21419285
- [Background] El Mubarak AH, Abu-bakr NH, Ibrahim YE. Postoperative pain in multiple-visit and single-visit root canal treatment. J Endod. 2010 Jan;36(1):36-9. doi: 10.1016/j.joen.2009.09.003. PMID 20003932
- [Background] Kovac J, Kovac D. Effect of irrigating solutions in endodontic therapy. Bratisl Lek Listy. 2011;112(7):410-5. PMID 21744739
- [Background] Saleh IM, Ruyter IE, Haapasalo M, Orstavik D. Survival of Enterococcus faecalis in infected dentinal tubules after root canal filling with different root canal sealers in vitro. Int Endod J. 2004 Mar;37(3):193-8. doi: 10.1111/j.0143-2885.2004.00785.x. PMID 15009409
- [Background] Estrela C, Estrela CR, Barbin EL, Spano JC, Marchesan MA, Pecora JD. Mechanism of action of sodium hypochlorite. Braz Dent J. 2002;13(2):113-7. doi: 10.1590/s0103-64402002000200007. PMID 12238801
- [Background] Siqueira JF Jr, Machado AG, Silveira RM, Lopes HP, de Uzeda M. Evaluation of the effectiveness of sodium hypochlorite used with three irrigation methods in the elimination of Enterococcus faecalis from the root canal, in vitro. Int Endod J. 1997 Jul;30(4):279-82. doi: 10.1046/j.1365-2591.1997.00096.x. PMID 9477814
- [Background] Siqueira JF Jr, Rocas IN, Favieri A, Lima KC. Chemomechanical reduction of the bacterial population in the root canal after instrumentation and irrigation with 1%, 2.5%, and 5.25% sodium hypochlorite. J Endod. 2000 Jun;26(6):331-4. doi: 10.1097/00004770-200006000-00006. PMID 11199749
- [Background] McComb D, Smith DC. A preliminary scanning electron microscopic study of root canals after endodontic procedures. J Endod. 1975 Jul;1(7):238-42. doi: 10.1016/S0099-2399(75)80226-3. No abstract available. PMID 1061799
- [Background] Grigoratos D, Knowles J, Ng YL, Gulabivala K. Effect of exposing dentine to sodium hypochlorite and calcium hydroxide on its flexural strength and elastic modulus. Int Endod J. 2001 Mar;34(2):113-9. doi: 10.1046/j.1365-2591.2001.00356.x. PMID 11307259
- [Background] Sim TP, Knowles JC, Ng YL, Shelton J, Gulabivala K. Effect of sodium hypochlorite on mechanical properties of dentine and tooth surface strain. Int Endod J. 2001 Mar;34(2):120-32. doi: 10.1046/j.1365-2591.2001.00357.x. PMID 11307260
- [Background] Mohammadi Z, Abbott PV. Antimicrobial substantivity of root canal irrigants and medicaments: a review. Aust Endod J. 2009 Dec;35(3):131-9. doi: 10.1111/j.1747-4477.2009.00164.x. PMID 19961451
- [Background] Torabinejad M, Cho Y, Khademi AA, Bakland LK, Shabahang S. The effect of various concentrations of sodium hypochlorite on the ability of MTAD to remove the smear layer. J Endod. 2003 Apr;29(4):233-9. doi: 10.1097/00004770-200304000-00001. PMID 12701769
- [Background] Shabahang S, Torabinejad M. Effect of MTAD on Enterococcus faecalis-contaminated root canals of extracted human teeth. J Endod. 2003 Sep;29(9):576-9. doi: 10.1097/00004770-200309000-00008. PMID 14503830
- [Background] Zhang W, Torabinejad M, Li Y. Evaluation of cytotoxicity of MTAD using the MTT-tetrazolium method. J Endod. 2003 Oct;29(10):654-7. doi: 10.1097/00004770-200310000-00010. PMID 14606789
- [Background] Machnick TK, Torabinejad M, Munoz CA, Shabahang S. Effect of MTAD on flexural strength and modulus of elasticity of dentin. J Endod. 2003 Nov;29(11):747-50. doi: 10.1097/00004770-200311000-00015. PMID 14651283
- [Background] Pinheiro ET, Gomes BP, Drucker DB, Zaia AA, Ferraz CC, Souza-Filho FJ. Antimicrobial susceptibility of Enterococcus faecalis isolated from canals of root filled teeth with periapical lesions. Int Endod J. 2004 Nov;37(11):756-63. doi: 10.1111/j.1365-2591.2004.00865.x. PMID 15479258
- [Background] Misuriya A, Bhardwaj A, Bhardwaj A, Aggrawal S, Kumar PP, Gajjarepu S. A comparative antimicrobial analysis of various root canal irrigating solutions on endodontic pathogens: an in vitro study. J Contemp Dent Pract. 2014 Mar 1;15(2):153-60. doi: 10.5005/jp-journals-10024-1506. PMID 25095835
- [Background] Shailaja S, Bhat SS, Hegde SK. Comparison between the antibacterial efficacies of three root canal irrigating solutions: antibiotic containing irrigant, Chlorhexidine and Chlorhexidine + Cetrimide. Oral Health Dent Manag. 2013 Dec;12(4):295-9. PMID 24390032
- [Background] Garlapati R, Venigalla BS, Surakanti JR, Thumu J, Chennamaneni KC, Kalluru RS. Comparison of the Antimicrobial Efficacy of Two Antibiotics Sparfloxacin and Augmentin as Experimental Root Canal Irrigating Solutions against Enterococcus faecalis - An Invitro Study. J Clin Diagn Res. 2016 Mar;10(3):ZC57-60. doi: 10.7860/JCDR/2016/17199.7470. Epub 2016 Mar 1. PMID 27135003
- [Background] Kamberi B, Bajrami D, Stavileci M, Omeragiq S, Dragidella F, Kocani F. The Antibacterial Efficacy of Biopure MTAD in Root Canal Contaminated with Enterococcus faecalis. ISRN Dent. 2012;2012:390526. doi: 10.5402/2012/390526. Epub 2012 Aug 1. PMID 22991671
- [Background] Agrawal V, Rao MR, Dhingra K, Gopal VR, Mohapatra A, Mohapatra A. An in vitro comparison of antimicrobial effcacy of three root canal irrigants-BioPure MTAD, 2% chlorhexidine gluconate and 5.25% sodium hypochlorite as a final rinse against E. faecalis. J Contemp Dent Pract. 2013 Sep 1;14(5):842-7. doi: 10.5005/jp-journals-10024-1413. PMID 24685785
- [Background] Mohammadi Z, Shalavi S, Giardino L, Palazzi F, Mashouf RY, Soltanian A. Antimicrobial effect of three new and two established root canal irrigation solutions. Gen Dent. 2012 Nov-Dec;60(6):534-7; quiz p.538-9. PMID 23220309
- [Background] Torabinejad M, Shabahang S, Bahjri K. Effect of MTAD on postoperative discomfort: a randomized clinical trial. J Endod. 2005 Mar;31(3):171-6. doi: 10.1097/01.don.0000137642.50944.a2. PMID 15735462
- [Background] Jain P, Yeluri R, Garg N, Mayall S, Rallan M, Gupta S, Pathivada L. A Comparative Evaluation of the Effectiveness of Three Different Irrigating Solution on Microorganisms in the Root Canal: An Invivo Study. J Clin Diagn Res. 2015 Dec;9(12):ZC39-42. doi: 10.7860/JCDR/2015/13133.6991. Epub 2015 Dec 1. PMID 26816990
- [Background] Tulsani SG, Chikkanarasaiah N, Bethur S. An in vivo comparison of antimicrobial efficacy of sodium hypochlorite and Biopure MTAD against enterococcus faecalis in primary teeth: A qPCR study. J Clin Pediatr Dent. 2014 Fall;39(1):30-4. doi: 10.17796/jcpd.39.1.c4q2155r16817219. PMID 25631723
- [Background] Siqueira JF Jr, Rocas IN, Favieri A, Machado AG, Gahyva SM, Oliveira JC, Abad EC. Incidence of postoperative pain after intracanal procedures based on an antimicrobial strategy. J Endod. 2002 Jun;28(6):457-60. doi: 10.1097/00004770-200206000-00010. PMID 12067129
- [Background] Almeida G, Marques E, De Martin AS, da Silveira Bueno CE, Nowakowski A, Cunha RS. Influence of irrigating solution on postoperative pain following single-visit endodontic treatment: randomized clinical trial. J Can Dent Assoc. 2012;78:c84. PMID 22985896